CLINICAL TRIAL: NCT02113150
Title: A Comparison of the Effects of Ketamine and Remifentanil on Serum Cystatin-c Levels in CABG Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turkiye Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, aslı demir, Z.Aslı Demir, MD, Assoc.Prof, Turkiye Yuksek Ihtisas Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TurkiyeYIH; Zaslidem (Registry Identifier: aslı demir)
Record Dates: First submitted 2014-03-23; First posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Coronary Artery Disease
Keywords: troponin t,cystatin-c,ketamine,remifentanil
MeSH Terms: conditions — Coronary Artery Disease | interventions — Remifentanil; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- remifentanil (Active Comparator): remifentanil, short acting opioid
  Interventions: Drug: Ketamine
- ketamine (Active Comparator): ketamine, intravenous anesthetic
  Interventions: Drug: remifentanil

INTERVENTIONS:
Drug: remifentanil — renal function
  Other Names: Ultiva
  Arms: ketamine
Drug: Ketamine — renal function
  Other Names: ketalar
  Arms: remifentanil

SUMMARY:
In this prospective, randomized, clinical trial, we have investigated the effects of ketamine-based and remifentanil-based anesthetic protocol on perioperative serum cystatin-c levels, and creatinine and/or cystatin-c based eGFR equations in terms of acute kidney injury in CABG surgery.This study was approved by the Ethics Committee of Hospital and all patients were informed and gave written consent. Patients scheduled for elective CABG with cardiopulmonary bypass. Patients were randomly allocated to anesthesia with remifentanil-propofol-midazolam (RPM) group or ketamine-propofol-midazolam (KPM) group. Blood samples were obtained before induction of anesthesia (baseline), at the end of the operation, and postoperative days 1, 2, and 4.

ELIGIBILITY:
Inclusion Criteria:

patients undergoing elective CABG with cardiopulmonary bypass

Exclusion Criteria:

patients undergoing emergency operation, combined operation, off-pump surgery, repeat surgery or valve surgery, patients presenting with chronic kidney disease or renal impairment, patients younger than 18 years old and neurological and/or psychiatric disturbances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-05; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
creatinin, BUN | 2 months

SECONDARY OUTCOMES:
Cystatin-c level | 2 months

OTHER OUTCOMES:
GFR value | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Aslı Demir, Principal Investigator — Turkey Yuksek Ihtisas Education and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Aslı Demir, Ankara, Ankara
  - Turkey Yuksek Ihtisas Education and Research Hospital, Ankara